CLINICAL TRIAL: NCT05246696
Title: Perceptions of Their Own Body and of the Body of Their Child Among Young Mothers With Anorexia Nervosa
Acronym: BodyBabe2
Status: Withdrawn | Type: Observational
Why Stopped: The project was to be led by midwives but the director of the school of midwives opposed it at the last moment...
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: RNI 2021 VILLEMEYRE-PLANE; 2021-A02824-37 (Other: 2021-A02824-37)
Record Dates: First submitted 2022-02-09; First posted 2022-02-18 (Actual); Last update posted 2022-10-19 (Actual); Status verified 2022-02

CONDITIONS: Anorexia Nervosa; Eating Disorders
Keywords: mother anorexia nervosa; body perception; post-partum; baby body
MeSH Terms: conditions — Anorexia Nervosa; Feeding and Eating Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient group
  Interventions: Other: BodyBabe questionnaire

INTERVENTIONS:
Other: BodyBabe questionnaire — assessment of young mothers' perceptions using self-questionnaires

SUMMARY:
The BodyBabe studies aims to evaluate the perceptions that young mothers with anorexia nervosa (active or in remission) have of their own body and of the body of their child. The evaluations are carried out with self-assessment questionnaires and silhouette scales at three time points: D0 (during the stay at the maternity hospital), D15 (15 days after delivery) and M9 (9 months after delivery).

The output expected from this study is to validate a questionnaire to help healthcare providers to adapt their care of women with anorexia nervosa during the pregnancy and the post-partum period.

DETAILED DESCRIPTION:
During the stay at maternity hospital, healthcare providers will identify potential candidates for the study on a daily basis according to the following criteria :

* BMI at the beginning of the pregnancy lower than 18,5 kg/m2 And/or
* History of anorexia nervosa

Tools and methods

The questionnaires used for the self-assessments are the following :

* Two questionnaires that evaluate the body satisfaction

  * The Body Shape Questionnaire (BSQ)
  * A questionnaire assessing the satisfaction of the mother regarding her baby's body shape (BodyBabe questionnaire).
* Two silhouette scales

  * Stunkard scale also called Figure Rating Scale (FRS)5
  * Infant Body Figure Drawings
* A questionnaire evaluating the severity of the eating disorders : Eating Attitude Test (EAT)
* A questionnaire detecting depression symptoms during post-partum : Edinburgh Post-natal Depression Scale (EPDS)

ELIGIBILITY:
Inclusion Criteria:

* adult woman, understanding and reading French, delivering in the CHU (Centre Hospitalier Universitaire) Clermont-Ferrand maternity hospital between 01/15/2020 and 01/14/2021, and with active or in remission anorexia nervosa diagnosed according to DSM-5 criteria (Diagnostic and Statistical Manual of Mental Disorders)
* able to accept participating to the study
* Affiliated to the national healthcare system

Exclusion Criteria:

* delivery before 32 weeks of amenorrhea (significant prematurity and extreme prematurity)
* death in utero or medically-motivated induced termination
* infant death during labour or post-partum
* refusal to participate

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: adult woman delivering in the CHU Clermont-Ferrand maternity hospital with active or in remission anorexia nervosa diagnosed according to DSM-5 criteria
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2022-06 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
evaluate the internal and external validity of the BodyBabe questionnaire | day1, day 15, day 270
  the internal validity of the questionnaire will be assessed with a factorial analysis. The internal consistency between sub-scales will be evaluated with the Cronbach α coefficient. The Spearman coefficient will be used to evaluate the item-subscale and inter-subscale correlation. The external validity will be estimated with Spearman correlation coefficient between different subscales. The reproducibility will be assessed by "test-request" at an interval of 15 days. Intra-class coefficients will be calculated for each subscale

SECONDARY OUTCOMES:
impact of the history of anorexia nervosa or severity on the questionnaires' scores | day1, day 15, day 270
  the scores will be compared to the state of the disease (active or in remission). Student Tests or ANOVA (non-parametric average comparisons from Mann-Whitney or Kruskal-Wallis for non-gaussian variables) will be implemented.

CONTACTS AND LOCATIONS:
Overall Officials: Michèle Villemeyre-Plane, Principal Investigator — University Hospital, Clermont-Ferrand